CLINICAL TRIAL: NCT00404781
Title: Pilot Study of Personal Optimized Antiplatelet Treatment After Percutaneous Coronary Intervention in Patients With Acute Coronary Syndromes
Brief Title: Effects of Optimized Antiplatelet Treatment After Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Yaling Han, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH-2006-C001
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Ischemic Heart Disease; Acute Coronary Syndromes
Keywords: ischemic heart disease; acute coronary syndromes; percutaneous transluminal coronary angioplasty; platelet function; aspirin; clopidogrel; cilostazol
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome | interventions — Cilostazol; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- optimal antiplatelet (Experimental): cilostazol in addition to aspirin and clopdidogrel for pts with clopidogrel resistance
  Interventions: Drug: cilostazol in addition to aspirin and clopidogrel
- standard antiplatelet (Active Comparator): aspirin and clopidogrel for all patients
  Interventions: Drug: cilostazol in addition to aspirin and clopidogrel

INTERVENTIONS:
Drug: cilostazol in addition to aspirin and clopidogrel

SUMMARY:
Effects of dual antiplatelet therapy with aspirin and clopidogrel after percutaneous coronary intervention has been proven. However, patients with low response to those agents are reported be associated with adverse clinical outcomes. We suppose that optimized antiplatelet therapy for individual patients based on platelet function assay may improve long-term outcomes especially in patients with high risk of thrombosis. In this prospective randomized study, patients in control group all receive standard dual antiplatelet therapy, and patients in optimized group receive different antiplatelet therapy according to risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* non-ST-segment elevated acute coronary syndromes
* patients undergoing selective or emergent PCI

Exclusion Criteria:

* administration of clopidogrel or ticlopidine within 2 weeks
* ST-segment elevated myocardial infarction
* contraindications of antiplatelet therapy
* history of intracranial bleeding
* known bleeding disorders
* severe liver or kidney disease

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events at 1 year | 1 year

SECONDARY OUTCOMES:
Hemorrhage events at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, M.D., Principal Investigator — Shenyang Northern Hospital
Locations (1):
- Northern Hospital, Shenyang, Liaoning, China